CLINICAL TRIAL: NCT03459742
Title: A Gamification Strategy to Reduce Childhood Obesity in Santiago Schools: a Cluster Randomized Controlled Trial
Brief Title: Juntos Santiago: Gamification Strategy to Reduce Childhood Obesity in Schools in Santiago de Chile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Municipality of Santiago (Other Government)
Collaborators: Delivery Associates (Unknown); Bloomberg Philanthropies (Other); University of Chile (Other); Pontificia Universidad Catolica de Chile (Other); Ministry of Health, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Secc. 2da. 11058
Record Dates: First submitted 2018-02-18; First posted 2018-03-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Obesity
Keywords: Obesity; Gamification; Schools; Cluster Randomized Trial
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial. The randomization unit will be the schools. The primary outcome will be measured individually, but the effect size will also be calculated at the school level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Gamification strategy. In 2018, the intervention group are 15 schools from Municipality of Santiago. In 2019, the intervention will cover all eligible schools in the Municipality of Santiago.
  Interventions: Behavioral: Gamification strategy
- Control (No Intervention): In 2018, the control group will be 5 randomly selected schools from Municipality of Santiago and 4 schools from Municipality of Estación Central. In 2019, the control group will be 4000 participants chosen from neighboring municipalities

INTERVENTIONS:
Behavioral: Gamification strategy — The intervention is a gamification strategy, including game elements such as points, levels and rewards. Points are scored by completion of healthy challenges, i.e. a healthy snacks challenge, a steps challenge and activity challenge. Intervention takes place for 8 months from Mar to Nov. There will be three levels. Level 1 at baseline, level 2 expected at month 4 by 100% of participants and level 3 expected in month 8 by 70% of participants. A new cycle will start in 2019.
  Rewards include an initial reward (Starting Kit), a structural reward and an activity reward. The Starting Kit is a box with souvenirs, information for students and teachers. A structural reward, at level 2, will be achieved collectively by all participating classes in one school. It consists of school infrastructure improvements to promote a healthy nutrition and PA (eg. climbing wall, shared bicycles, sports equipment). An activity reward (AR), when reaching level 3, consists of a fun and healthy activity.
  Arms: Intervention

SUMMARY:
School-based interventions have shown mixed results. Most studies have lacked enough statistical power and have been carried out in North America and Europe.

The Juntos Santiago is a cluster-randomized trial based on a gamification strategy conducted in Santiago de Chile. The trial uses elements of a game such as points, levels and rewards along with a strong community participation component.

Children voted their enrollment and collectively chose the rewards (two per year, one activity and another structural) they are playing for. The intervention consists of a healthy snacks challenge, a steps challenge and an activity challenge. The primary outcome is change in z-BMI and waist circumference.

DETAILED DESCRIPTION:
Purpose

Childhood obesity has reached epidemic proportions in the last decades. The growing obesity epidemic has negative health, economic and social consequences (Wang et al., 2011, Withrow and Alter, 2011, Griffiths et al., 2010). These include an increased risk of type 2 diabetes, cardiovascular diseases and cancer, a shorter life expectancy and lower quality of life (Wang et al., 2011, Olshansky et al., 2005). Studies suggest obese and physically inactive kids also have lower academic achievement (Correa-Burrows et al., 2016, Garcia-Hermoso and Marina, 2017).

The school environment is a suitable setting for implementing evidence-based interventions to reduce obesity. Several systematic reviews of RCTs have shown a modest decrease in adiposity and blood pressure (Oosterhoff et al., 2016, Wang et al., 2015, Sobol-Goldberg et al., 2013, Mei et al., 2016, Vasques et al., 2014). Oosterhoff et al (2016) showed a significant reduction in BMI of 0.22 kg/mt2 and systolic blood pressure, while no effect was found for diastolic blood pressure (Oosterhoff et al., 2016).

Multicomponent interventions addressing both nutrition and physical activity and involving parents and the school community have shown to be more effective (Wang et al., 2015). Few studies, however, have used a structured motivational strategy to increase engagement of students and school communities.

The clustered-randomized controlled trial Juntos Santiago was designed as a multidimensional intervention that incorporates a gamification strategy to increase motivation and participation. The intervention addresses the snacks brought from home, encourages physical activity and active parent and school community participation. All the aspects of the intervention are brought together in a game that provides points, levels and rewards that improve school infrastructure for better nutrition and physical activity. Structural rewards contribute to a sustained effect of the intervention.

The purpose of the Juntos Santiago study is to examine the effectiveness of a multicomponent school-based gamification strategy to reduce the body mass index (BMI), waist circumference (WC) and systolic blood pressure (SBP) in school children in 5th and 6th grade, compared to usual care and a leaflet and designed to prevent obesity.

Intervention

The study is part of the Juntos Santiago project, which will be progressively scaled-up for three years. A pilot will be carried out in three schools during 2017, without a control group. In 2018, the trial will include 12 randomly selected schools; the control group will be randomly selected from schools in the Municipality of Santiago plus 4 schools in a neighbour municipality (Estación Central). In 2019, the trial will expand to include all eligible schools in the Municipality of Santiago and 4000 students in the control group from neighbouring municipalities.

The intervention is based on the socio-ecological model. The intervention is a gamification strategy consisting of four components:

Gamification incentives, including the use of points, levels and rewards, to promote behavioural and structural change in the schools. The gamification strategy bundles the intervention components together.

Healthy challenges. Children will be invited to participate in healthy challenges. They will score points, which will result in progressing into a next level and win rewards at the end of the year. There will be three types of challenges:

Healthy snacks challenge, where children collect points for bringing healthy snacks for school breaks.

Steps challenge, where children and one caretaker are given an activity tracker three times a year for two weeks. Points are collected each time a child or a caretaker surpasses a daily threshold level Activity challenge, where children and their families collect points by uploading pictures of specific healthy activities defined by the research team.

Levels. The intervention will take place throughout the year (8 months from March to November). There will be three levels, each associated with a specific reward. Level 1 is the starting point. Level 2 is planned to be reached by 100% at 4 months of the intervention. Level 3 is planned be reached by 70% towards the end of the intervention year. A new cycle will start in 2019.

Rewards. The intervention includes the following rewards:

An initial reward (Starting Kit). The Starting Kit is a box that includes project souvenirs for students, guidelines on healthy snacks and physical activity for children and their families and 12 teaching modules on healthy behaviours designed for teachers. The Starting Kit is delivered upon enrolment in the trial.

An structural reward (SR) when reaching level 2. This reward will be achieved collectively by all participating classes in one school. The reward will be selected from a closed list and will consist of improvements of the school infrastructure to promote a healthy nutrition and physical activity (e.g. a school garden, playground facilities, climbing wall, shared bicycles, sports equipment).

An activity reward (AR) when reaching level 3. This reward will be achieved by each class and will consist of a fun and healthy activity. For example, the visit of a famous sport player, an outdoor trip, tickets to an amusement park, etc.

Parental involvement. Parents will be involved indirectly by the healthy snacks and directly in the steps and activity challenges. Parents will receive a SMS each time points are awarded.

A web platform will be developed for schools and classes to track progress of their points, levels and rewards. An individual login by each student will allow the student and their families to check the results of the anthropometric measurements and points awarded.

Measurements Intervention measurement Healthy snacks. Healthy snacks will be measured three times per month by a trained team. In packaged snacks, data will be collected using the stock keeping unit (SKU) in the barcode. Non-packaged foods will be divided into predefined categories. A food composition database including the calories, saturated fats, total sugar and salt per 100 grams has been developed for this purpose. Indicators: Mean change in calories, saturated fat, total sugar and salt per 100 grams.

Steps challenge. Steps will be measured using a validated activity tracker for 14 days. The mean daily steps will be measured. Indicator: Mean change in total daily steps.

Activity challenge. The research team will define activities were children and families who complete these activity challenges will collect points. This include activities organized by the Municipality of Santiago (i.e. a City run), healthy activities to do as a family (such as cycling or walking together or having a healthy lunch following predefined guidelines), and class activities organized by the teacher following also predefined guidelines. Students and their families will upload pictures of these activities to the web platform to collect the points. A validation system Given the All uploaded pictures Indicator: Mean change in number of completed activity challenges.

Intermediate variables A self-administered questionnaire will be applied at baseline and month 8. The questionnaire includes validated instruments to assess consumption of fruits and vegetables, unhealthy snacks and moderate and vigorous physical activity (MVPA). Consumption of food and vegetables and unhealthy snacks will be measured using the instrument validated by Lera et al (2015) developed in Chilean children aged 10 to 11 years old.12 Additionally, questions from the Global School Health Survey 2013 developed jointly by the Centre for Disease Prevention (CDC) and the Ministry of Health (MoH).

Physical activity will be measured using the PAQ-C. PAQ-C has shown high validity and reliability in different settings. The study will use the PAQ-C version implemented in Chilean schools by Zuñiga et al (2017).13 Questions from the GSHS 2013 on physical activity will also be included.

Adverse effects The study will monitor the experience of bullying, as a possible adverse effect of the intervention, using two questions from the GSHS 2013 on the frequency of bullying in the past 30 days and type of bullying.

ELIGIBILITY:
Inclusion Criteria:

* Students in schools in Santiago in 5th and 6th grade (approximately 10 and 11 years old)
* Willingness to participate in the intervention and measurements
* Able to read Spanish and accurately complete dietary assessments
* Any weight status

Exclusion Criteria:

* School not accepting to participate in the study
* Class votes against enrolling in the study
* Caretaker does not grant permission to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in zBMI | Measured at baseline and 8 months
  Change in zscore of body mass index at 8 months
Change in waist circumference | Measured at baseline and 8 months
  Change in waist circumference measured using standard protocols at 8 months

SECONDARY OUTCOMES:
Change in BMI | Measured at baseline and 8 months
  Change in body mass index (weight/height squared) at 8 months. Weight and height will be combined to report BMI in kg/m^2
Change in SBP | Measured at baseline and 8 months
  Change in systolic blood pressure at 8 months
Change in DBP | Measured at baseline and 8 months
  Change in diastolic blood pressure at 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Peña, MD, MSc, Study Chair — Finnish Institute for Health and Welfare; Macarena Carranza, LDN, MSc, Principal Investigator — Municipality of Santiago; Pedro Zitko, MD, MSc, Study Chair — King's College London
Locations (2):
- Chile (2):
  - Estacion Central, Santiago, N/A = Not Applicable
  - Santiago, Santiago, N/A = Not Applicable

IPD SHARING:
Plan to Share IPD: Undecided
Data without unique personal identification number will be available to associated researchers

REFERENCES:
- [Background] Wang YC, McPherson K, Marsh T, Gortmaker SL, Brown M. Health and economic burden of the projected obesity trends in the USA and the UK. Lancet. 2011 Aug 27;378(9793):815-25. doi: 10.1016/S0140-6736(11)60814-3. PMID 21872750
- [Background] Withrow D, Alter DA. The economic burden of obesity worldwide: a systematic review of the direct costs of obesity. Obes Rev. 2011 Feb;12(2):131-41. doi: 10.1111/j.1467-789X.2009.00712.x. PMID 20122135
- [Background] Griffiths LJ, Parsons TJ, Hill AJ. Self-esteem and quality of life in obese children and adolescents: a systematic review. Int J Pediatr Obes. 2010 Aug;5(4):282-304. doi: 10.3109/17477160903473697. PMID 20210677
- [Background] Olshansky SJ, Passaro DJ, Hershow RC, Layden J, Carnes BA, Brody J, Hayflick L, Butler RN, Allison DB, Ludwig DS. A potential decline in life expectancy in the United States in the 21st century. N Engl J Med. 2005 Mar 17;352(11):1138-45. doi: 10.1056/NEJMsr043743. PMID 15784668
- [Background] Correa-Burrows P, Burrows R, Blanco E, Reyes M, Gahagan S. Nutritional quality of diet and academic performance in Chilean students. Bull World Health Organ. 2016 Mar 1;94(3):185-92. doi: 10.2471/BLT.15.161315. Epub 2016 Feb 3. PMID 26966329
- [Background] Garcia-Hermoso A, Marina R. Relationship of weight status, physical activity and screen time with academic achievement in adolescents. Obes Res Clin Pract. 2017 Jan-Feb;11(1):44-50. doi: 10.1016/j.orcp.2015.07.006. Epub 2015 Aug 3. PMID 26249128
- [Background] Oosterhoff M, Joore M, Ferreira I. The effects of school-based lifestyle interventions on body mass index and blood pressure: a multivariate multilevel meta-analysis of randomized controlled trials. Obes Rev. 2016 Nov;17(11):1131-1153. doi: 10.1111/obr.12446. Epub 2016 Jul 19. PMID 27432468
- [Background] Wang Y, Cai L, Wu Y, Wilson RF, Weston C, Fawole O, Bleich SN, Cheskin LJ, Showell NN, Lau BD, Chiu DT, Zhang A, Segal J. What childhood obesity prevention programmes work? A systematic review and meta-analysis. Obes Rev. 2015 Jul;16(7):547-65. doi: 10.1111/obr.12277. Epub 2015 Apr 20. PMID 25893796
- [Background] Sobol-Goldberg S, Rabinowitz J, Gross R. School-based obesity prevention programs: a meta-analysis of randomized controlled trials. Obesity (Silver Spring). 2013 Dec;21(12):2422-8. doi: 10.1002/oby.20515. Epub 2013 Aug 13. PMID 23794226
- [Background] Mei H, Xiong Y, Xie S, Guo S, Li Y, Guo B, Zhang J. The impact of long-term school-based physical activity interventions on body mass index of primary school children - a meta-analysis of randomized controlled trials. BMC Public Health. 2016 Mar 1;16:205. doi: 10.1186/s12889-016-2829-z. PMID 26931236
- [Background] Vasques C, Magalhaes P, Cortinhas A, Mota P, Leitao J, Lopes VP. Effects of intervention programs on child and adolescent BMI: A meta-analysis study. J Phys Act Health. 2014 Feb;11(2):426-44. doi: 10.1123/jpah.2012-0035. Epub 2013 Jan 30. PMID 23363556
- [Background] Lera L, Fretes G, Gonzalez CG, Salinas J, Vio del Rio F. [Validity of an instrument for assessing food consumption, food habits and cooking skills in 8-11 years old students]. Nutr Hosp. 2015 May 1;31(5):1977-88. doi: 10.3305/nh.2015.31.5.8607. Spanish. PMID 25929365
- [Background] Zurita-Ortega F, Castro-Sanchez M, Rodriguez-Fernandez S, Cofre-Bolados C, Chacon-Cuberos R, Martinez-Martinez A, Muros-Molina JJ. [Physical activity, obesity and self-esteem in chilean schoolchildren]. Rev Med Chil. 2017 Mar;145(3):299-308. doi: 10.4067/S0034-98872017000300006. Spanish. PMID 28548189